CLINICAL TRIAL: NCT04545567
Title: Fully Automated Closed Loop Control in Adolescents With Type 1 Diabetes (Rocket AP)
Brief Title: Fully Automated Closed Loop Control in Adolescents With Type 1 Diabetes
Acronym: RocketAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Mark D. DeBoer, MD, MSc., MCR, Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 200235
Record Dates: First submitted 2020-09-03; First posted 2020-09-11 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes
Keywords: Artificial Pancreas (AP); Continuous Glucose Monitor (CGM); Insulin Pump; Closed Loop Control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: A randomized cross-over trial assessing glycemic responses to two different approaches to insulin dosing for carbohydrate ingestion (announced vs. unannounced), with two different AP systems (RocketAP vs. USS Virginia, aka Control-IQ, in random order)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- RocketAP (Experimental): Adolescents will be assessed for a 48-70 hour period on the Rocket AP. This time will include two dinner times, one with and one without announcement of carbohydrate content. This is a cross-over study, so all participants will also be tested on the USS Virginia system under the same conditions.
  Interventions: Device: RocketAP
- USS Virginia (Active Comparator): Adolescents will be assessed for a 48-70 hour period on the USS Virginia system. This time will include two dinner times, one with and one without announcement of carbohydrate content. This is a cross-over study, so all participants will also be tested on the Rocket AP system under the same conditions.
  Interventions: Device: USS Virginia

INTERVENTIONS:
Device: RocketAP — Artificial pancreas system which is designed to be able to identify when you have eaten and provide insulin for this meal
  Arms: RocketAP
Device: USS Virginia — Artificial pancreas system which responds to glucose fluctuations by modulating insulin delivery but does not specifically detect meal ingestion
  Arms: USS Virginia

SUMMARY:
The study team will be comparing two investigational Artificial Pancreas (AP) systems that the UVA Center for Diabetes Technology has developed. An artificial pancreas system delivers insulin automatically based on a blood glucose level that is provided from a continuous glucose monitor (CGM).

DETAILED DESCRIPTION:
Maintaining blood glucose (BG) control among adolescents with Type 1 diabetes (T1D) is arguably the greatest challenge in the entire field of T1D. One reason for this poor control relates to missed meal boluses, which affects 65% of adolescents at least once weekly, with 38% missing at least 15% of their boluses. Adolescents who miss four boluses weekly experience an increase of 1% in their HbA1c. While the advent of the artificial pancreas (AP) offers promise of safe reductions in HbA1c, the study team previously found that the AP only partly compensates for missed prandial insulin -demonstrating that some form of meal announcement is necessary for good BG control, even with an AP. One way to automate this process is by sharing the prandial dosing responsibilities between an automated insulin priming (based on continuous glucose monitor condition predictive of a safe situation for such insulin dosing) and a closed loop controller capable of reconstructing (estimating) the prevailing glucose rate of appearance from an unannounced meal. The study team has developed such an insulin priming schema and integrated it into a new version of the robust Model Predictive Controller University of Virginia AP system (called the RocketAP).

In the current study, the investigators are testing this new AP system in two configurations: hybrid and fully automated, among up to 20 adolescents. The primary outcome will be one of efficacy in assessing how well the new system controls post-prandial BG in the absence of carbohydrate (CHO) announcement as compared to the same situation but using the Control-IQ closed loop algorithm, also designed at UVa and using the same modular architecture and safety system, but without insulin priming and with a less advanced model-based controller. Further comparisons will be made to BG control on RocketAP with CHO announcement and on Control-IQ with CHO announcement. Adolescents will be started on the respective University of Virginia AP systems (RocketAP and Control-IQ in random order, both implemented on the DiAs platform, MAF 2109) and followed over the course of two dinners on each of the two platforms: a dinner where CHO is announced as normal and the 2nd where no announcement is made.

The study team hypothesize that performances of RocketAP in fully automated mode will lie in between Hybrid and Fully Automated Control-IQ. In time, this may provide an opportunity to improve BG control among adolescents who miss meal announcement.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥12.0 and ≤25 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
3. Currently using insulin for at least six months
4. Currently using insulin pump for at least three months
5. Using insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
6. Access to internet and willingness to upload data during the study as needed
7. For females, not currently known to be pregnant or breastfeeding
8. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
9. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use
10. Willingness to use the UVa artificial pancreas system throughout study sessions.
11. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study
12. Total daily insulin dose (TDD) at least 10 U/day and not more than 100 U/d
13. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, biguanides, sulfonylureas and naturaceuticals)
14. Willingness to eat at least 1 g/kg of carbohydrate per day during the camp/hotel admission
15. Willingness to reschedule Study Dinner Sessions if placed on oral steroids
16. An understanding and willingness to follow the protocol and signed informed consent

Exclusion Criteria:

1. History of diabetic ketoacidosis (DKA) in the 12 months prior to enrollment
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
3. Pregnancy or intent to become pregnant during the trial
4. Currently being treated for a seizure disorder
5. Planned surgery during study duration
6. Treatment with any non-insulin glucose-lowering agent (including metformin, GLP-1 agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals)
7. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
8. Use of an automated insulin delivery mechanism that is not downloadable by the subject or study team

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D DeBoer, MD, MSc, MCR, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Pending
Supporting Information: Study Protocol, ICF
Time Frame: Generally will be available after publications completed.
Access Criteria: No restrictions for access.

REFERENCES:
- [Result] Garcia-Tirado J, Diaz JL, Esquivel-Zuniga R, Koravi CLK, Corbett JP, Dawson M, Wakeman C, Barnett CL, Oliveri MC, Myers H, Krauthause K, Breton MD, DeBoer MD. Advanced Closed-Loop Control System Improves Postprandial Glycemic Control Compared With a Hybrid Closed-Loop System Following Unannounced Meal. Diabetes Care. 2021 Aug 15:dc210932. doi: 10.2337/dc21-0932. Online ahead of print. PMID 34400480

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 subjects were recruited from October 2020 to mid-December 2020 either in person (UVA CDT facility) or by video conference.
Pre-assignment Details: Following study enrollment, participants were trained in the study devices. This study visit was followed by 4 weeks of CGM and pump data collection at the participant's home/usual routine. From the 21 enrolled participants, 1 did not follow up and 2 tested positive for SARS-co-V2 and were excluded from the study.
Groups:
- RocketAP First, Then USS Virginia: Participants were randomized following the Data Collection Phase in a 1:1 ratio. Participants in the Experimental-Control Arm underwent the Experimental Admission first, utilizing a meal-related fully automated artificial pancreas (AP) controller (RocketAP), followed by the Control Admission, which utilized a hybrid AP controller (USS-Virginia) with no washout period in between.
  During the 96-hour admission, study participants started using RocketAP (48h) around midday on Day 1 and switched to USS Virginia (48h) at midday on Day 3. Every 48-hour part of the admission consisted of quiet activities during the morning, lunch at 13:00, light walk at 17:00, dinner at 18:00, and quiet activities during the evening. Days 2 and 4 differed from Days 1 and 3, respectively, by the dinner announcements, i.e., dinner was not announced over Days 1 and 3 and was announced over Days 2 and 4.
- USS Virginia First, Then Rocket AP: Participants were randomized following the Data Collection Phase in a 1:1 ratio. Participants in the Control-Experimental Arm underwent the Control Admission first, utilizing a hybrid AP controller (USS-Virginia) first followed by a meal-related fully automated artificial pancreas (AP) controller (RocketAP) with no washout period in between.
  During the 96-hour admission, study participants started with USS Virginia (48h) around midday on Day 1 and switched to RocketAP (48h) at midday on Day 3. Every 48-hour part of the admission consisted of quiet activities during the morning, lunch at 13:00, light walk at 17:00, dinner at 18:00, and quiet activities during the evening. Days 2 and 4 differed from Days 1 and 3, respectively, by the dinner announcements, i.e., dinner was not announced over Days 1 and 3 and was announced over Days 2 and 4.
Period: Overall Study
Arm/Group | RocketAP First, Then USS Virginia | USS Virginia First, Then Rocket AP
Started | 10 | 11
Completed | 9 | 9
Not Completed | 1 | 2
Not completed — tested positive for SARS-co-V2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RocketAP First, Then USS Virginia | USS Virginia First, Then Rocket AP | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 8 | 17
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.4) | 16 (2) | 16 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 36
HbA1c [Mean (Standard Deviation); unit: % of HbA1c] | 7.7 (2) | 7.3 (1) | 7.4 (1.5)
Weight [Mean (Standard Deviation); unit: kg] | 65.2 (11.5) | 65.2 (11.5) | 65.2 (11.5)
Height [Mean (Standard Deviation); unit: cm] | 167 (9) | 167 (9) | 167 (9)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 7.7 (3.2) | 7.7 (3.2) | 7.7 (3.2)
Total daily insulin [Mean (Standard Deviation); unit: IU] | 60 (16.3) | 60 (16.3) | 60 (16.3)
Carbohydrate ratio [Mean (Standard Deviation); unit: g CHO per IU of insulin] — Insulin-to-carb ratio (ICR), also known as carbohydrate ratio (CR) or carbohydrate factor, is a calculation used to determine how many grams of carbs are covered by one unit of rapid-acting insulin for a person with diabetes.
  g CHO per IU of insulin | 7.7 (1.9) | 7.7 (1.9) | 7.7 (1.9)
Correction factor [Mean (Standard Deviation); unit: mg/dL glucose per IU insulin] — A Correction Factor (sometimes called insulin sensitivity), is how much 1 unit of rapid-acting insulin will generally lower the blood glucose (in mg/dL) of a given insulin-dependent person with diabetes.
  mg/dL glucose per IU insulin | 43 (18) | 43 (18) | 43 (18)
basal rate profile [Mean (Standard Deviation); unit: IU/h] — The basal rate is the amount of insulin per unit of time (h) that a given insulin-dependent person with diabetes needs to cover non-meal needs. Over a 24-hour period, the basal flow of insulin accounts for about 50% of a person's total daily insulin requirement.
  IU/h | 1.3 (0.4) | 1.3 (0.4) | 1.3 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time From Dinner Time Until Midnight With Blood Glucose in Range 70-180 mg/dL in the Unannounced Meal
Description: Percentage of time from dinner time until midnight with blood glucose in range 70-180 mg/dL in the unannounced meal
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: %Time in Range (TIR)
Groups:
- RocketAP: Adolescents will be assessed for a 48-hour period on Rocket AP (Experimental condition). This study portion included two dinners over two consecutive days, one with and one without timing/carbohydrate content announcement.
- USS Virginia: Adolescents will be assessed for a 48-hour period on USS Virginia (Control condition). This study portion included two dinners over two consecutive days, one with and one without timing/carbohydrate content announcement.
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
%Time in Range (TIR) | 83 [64 to 93] | 53 [40 to 71]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Hypoglycemia Events From Dinner Time Until Midnight
Description: Number of hypoglycemia events from dinner time until midnight
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: hypoglycemic event
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
hypoglycemic event | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Time From Dinner Time Until Midnight With Blood Glucose in Range < 70 mg/dL
Description: Percentage of Time From Dinner Time Until Midnight With Blood Glucose in Range < 70 mg/dL
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: % time<70mg/dL
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
% time<70mg/dL | 0 [0 to 1] | 0 [0 to 0]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.2, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage of Time From Dinner Time Until Midnight With Blood Glucose in Range >180 mg/dL
Description: Percentage of Time From Dinner Time Until Midnight With Blood Glucose in Range >180 mg/dL
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: % time>180mg/dL
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
% time>180mg/dL | 17 [1.3 to 34] | 47 [28 to 60]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percentage of Time From Dinner Time Until Midnight With Blood Glucose in Range >250 mg/dL
Description: Percentage of Time From Dinner Time Until Midnight With Blood Glucose in Range >250 mg/dL
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: % time>250mg/dL
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
% time>250mg/dL | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Units of Insulin Injected From Dinner Time Until Midnight
Description: Units of insulin injected from dinner time until midnight
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: IU of insulin
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
IU of insulin | 15 (5) | 14 (4)
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.21, t-test, 2 sided

7. Secondary Outcome: The Blood Glucose Area Under the Curve (AUC) From Dinner Until Midnight, Accounting for the Initial Blood Glucose Value
Description: The blood glucose area under the curve (AUC) from dinner until midnight, accounting for the initial blood glucose value.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: mg/dL * min
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
mg/dL * min | 27052 (1248) | 25840 (8134)
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.73

8. Secondary Outcome: Percentage of Time From Dinner Time Until Dinner Time + 12h With Blood Glucose in Range 70-180 mg/dL
Description: Percentage of time from dinner time until dinner time + 12h with blood glucose in range 70-180 mg/dL
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: %Time in Range (TIR)
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
%Time in Range (TIR) | 90 [79 to 96] | 75 [58 to 83]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Number of Hypoglycemia Events From Dinner Time Until Dinner Time + 12h
Description: Number of hypoglycemia events from dinner Time until dinner time + 12h
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: hypoglycemic event
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
hypoglycemic event | 0 [0 to 0.7] | 0 [0 to 1]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Percentage of Time From Dinner Time Until Dinner Time + 12h With Blood Glucose in Range <70 mg/dL
Description: Percentage of time from dinner time until dinner time + 12h with blood Glucose in range <70 mg/dL
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: % time<70mg/dL
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
% time<70mg/dL | 0 [0 to 1.2] | 0 [0 to 0.7]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Percentage of Time From Dinner Time Until Dinner Time + 12h With Blood Glucose >180 mg/dL
Description: Percentage of Time From Dinner Time Until Dinner Time + 12h With Blood Glucose >180 mg/dL
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: % time>180mg/dL
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
% time>180mg/dL | 8.7 [3 to 17] | 25 [14 to 37]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Percentage of Time From Dinner Time Until Dinner Time + 12h With Blood Glucose >250 mg/dL
Description: Percentage of Time From Dinner Time Until Dinner Time + 12h With Blood Glucose >250 mg/dL
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: % time>250mg/dL
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
% time>250mg/dL | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Units of Insulin Injected From Dinner Time Until Dinner Time + 12h
Description: Units of insulin injected from dinner time until dinner time + 12h
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
IU | 21 (8) | 20 (4)
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.28, t-test, 2 sided

14. Secondary Outcome: The Blood Glucose Area Under the Curve (AUC) From Dinner Until Dinner + 12h, Accounting for the Initial Blood Glucose Value
Description: The Blood Glucose Area Under the Curve (AUC) From Dinner Until dinner + 12h, Accounting for the Initial Blood Glucose Value
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: mg/dL * min
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
mg/dL * min | 38891 (16054) | 40671 (18110)
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.05, t-test, 1 sided; Mean Difference (Final Values) = 0.38

15. Secondary Outcome: Percentage of Time Outside the Dinner Sessions With Blood Glucose in Range 70-180 mg/dL
Description: Percentage of Time outside the dinner sessions With Blood Glucose in Range 70-180 mg/dL
Time Frame: 36 hours
Measure: Median (Inter-Quartile Range); unit: %Time in Range (TIR)
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
%Time in Range (TIR) | 86 [82 to 92] | 81 [76 to 86]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Number of Hypoglycemia Events Outside of the Study Dinner Sessions
Description: Number of hypoglycemia events outside of the Study Dinner Sessions
Time Frame: 36 hours
Measure: Median (Inter-Quartile Range); unit: hypoglycemic event
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
hypoglycemic event | 3 [1 to 5] | 4.5 [1 to 8]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.14, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Percentage of Time Outside of the Study Dinner Sessions With Blood Glucose <70 mg/dL
Description: Percentage of Time outside of the Study Dinner Sessions with Blood Glucose <70 mg/dL
Time Frame: 36 hours
Measure: Median (Inter-Quartile Range); unit: % time<70mg/dL
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
% time<70mg/dL | 2.2 [1 to 3.6] | 2.9 [0.9 to 4.8]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Other; p = 0.22, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Percent of Time Outside of the Study Dinner Sessions With Blood Glucose >180 mg/dL
Description: Percent of Time Outside of the Study Dinner Sessions with Blood Glucose >180 mg/dL
Time Frame: 36 hours
Measure: Median (Inter-Quartile Range); unit: % time>180mg/dL
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
% time>180mg/dL | 9.5 [5 to 13] | 14 [7 to 18]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Percent Time Outside of the Study Dinner Sessions With Blood Glucose >250 mg/dL
Description: Percent Time Outside of the Study Dinner Sessions with Blood Glucose >250 mg/dL
Time Frame: 36 hours
Measure: Median (Inter-Quartile Range); unit: % time>250mg/dL
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
% time>250mg/dL | 0 [0 to 1] | 0 [0 to 1.5]
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Units of Insulin Injected Outside of the Study Dinner Sessions
Description: Units of insulin injected outside of the Study Dinner Sessions
Time Frame: 36 hours
Measure: Mean (Standard Deviation); unit: IU of insulin
Arm/Group | RocketAP | USS Virginia
Number analyzed (Participants) | 18 | 18
IU of insulin | 78 (23) | 85 (20)
Statistical Analysis 1: Comparison: RocketAP vs USS Virginia; Test type: Superiority; p = 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 46h
Description: nothing to disclose in this field
Arm/Group | RocketAP | USS Virginia
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT04545567/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT04545567/ICF_001.pdf